CLINICAL TRIAL: NCT03638505
Title: Cross-sectional Study of the Factors Determining the Quality of Life of the Patient and the Burden of the Caregiver in Progressive Supranuclear Palsy
Brief Title: Quality of Life of the Patient and the Burden of the Caregiver in Progressive Supranuclear Palsy
Acronym: Qual-PSP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-62
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: patients with Progressive supranuclear palsy. PSP-QoL will be performed in this group
  Interventions: Other: PSP-QoL
- caregiver: the caregiver of the patient with Progressive supranuclear palsy PSP-QoL will be performed in this group
  Interventions: Other: PSP-QoL

INTERVENTIONS:
Other: PSP-QoL — PSP-QoL is a patient-reported outcome measure for progressive supranuclear palsy (PSP). The Supranuclear Palsy Quality of Life scale (PSP-QoL) may be a helpful patient-reported scale for clinical trials and studies in PSP.
  PSP-QoL consists of 28 items scored on a 3- or 5-point Likert scale, with the total score ranging from 0 to 100. Each item is scored from either 0 to 4, with the exception of four items, which are scored from 0 to 2, with higher scores indicating more-severe disability or movement abnormality. Items are in six categories: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. The scale includes comments and/or instructions for each item and word anchors to explain the ratings.

SUMMARY:
Progressive supranuclear palsy (PSP) is a rare neurodegenerative disease from the parkinsonian syndrome group.

PSP is characterised by the association of a non-doparesponsive parkinsonian syndrome with axial signs. The latter predominantly manifest as a psycho-motor slowness, an apathy and frontal executive deficits. Swallowing impairments may additionally provoke life-threatening situations. Today the treatment is mostly symptomatic as no cure is available. Given the limited treatment options and its clinical characteristics, PSP deeply impact on the patients' quality of life (QoL) as well as on their caregivers'. Nevertheless a limited number of studies have focused on these aspects. A better understaning of the factors determining both patient and cargiver QoL may help optimising their care.

the principal objective of this study is to identify the determinants of PSP patients' QoL.

The secondary objectives are : i) to identify the determinants (medical, behavioural, socio-economic, environmental …) of PSP patients' caregivers' QoL and burden ; ii) to validate in French language the QoL scale specific for PSP available in English (PSP-QoL).

This is a multidisciplinary transversal study. 2 subject groups will be included : i) PSP patients ; ii) caregiver of PSP patients (designated by the patient as being the person closest to them), Data collected : i) from the patient : socio-demographic, social and professionnal environment, clinical (disease duration and severity, neuropsychological evaluation), therapeutic, mood, anxiety, coping, body image, QoL ; ii) from the caregiver: socio-demographic, social and professionnal environment, connection with the patient, data relative to their own health, mood, anxiety, coping, QoL, burden.

Progress : patient information, designation of a caregiver, consent collection, collection of data Statistical analysis : To address the principal objective 'patient' QoL scores will be confronted to the other collected variables (Student's t-test, correlation coefficient). The results will be adjusted to the confounding factors using multivariate analyses.

DETAILED DESCRIPTION:
Progressive supranuclear palsy (PSP) is a rare neurodegenerative disease from the parkinsonian syndrome group. It represents 5 to 10% of all parkinsonian syndromes and affects 3000 to 10000 persons in France.

PSP is characterised by the association of a non-doparesponsive parkinsonian syndrome with axial signs such as early gait instability and falls, oculomotor signs such as a vertical gaze limitation and both cognitive and behavioural disturbances. The latter predominantly manifest as a psycho-motor slowness, an apathy and frontal executive deficits. Swallowing impairments may additionally provoke life-threatening situations. Today the treatment is mostly symptomatic as no cure is available. Given the limited treatment options and its clinical characteristics, PSP deeply impact on the patients' quality of life (QoL) as well as on their caregivers'. Nevertheless a limited number of studies have focused on these aspects. A better understaning of the factors determining both patient and cargiver QoL may help optimising their care.

Objectives : the principal objective of this study is to identify the determinants (motor, behavioural, socio-economic, environemental…) of PSP patients' QoL.

The secondary objectives are : i) to identify the determinants (medical, behavioural, socio-economic, environmental …) of PSP patients' caregivers' QoL and burden ; ii) to validate in French language the QoL scale specific for PSP available in English (PSP-QoL).

Methods : This is a multidisciplinary transversal study. Population : 2 subject groups will be included : i) PSP patients ; ii) caregiver of PSP patients (designated by the patient as being the person closest to them), Data collected : i) from the patient : socio-demographic, social and professionnal environment, clinical (disease duration and severity, neuropsychological evaluation), therapeutic, mood, anxiety, coping, body image, QoL ; ii) from the caregiver: socio-demographic, social and professionnal environment, connection with the patient, data relative to their own health, mood, anxiety, coping, QoL, burden.

Progress : patient information, designation of a caregiver, consent collection, collection of data Statistical analysis : To address the principal objective 'patient' QoL scores will be confronted to the other collected variables (Student's t-test, correlation coefficient). The results will be adjusted to the confounding factors using multivariate analyses. To address the secondary objective, 'caregiver' QoL and burden scores will be confronted to the other collected variables through the same procedure. The transcultural validation of the PSP-QoL scale will be obtained using standard methodology: forward-backward method, acceptability test, study of metric properties.

Expected results and impact: This work will help understanding the social handicap in PSP and may lead to new therapeutic strategies.

Relevance of the project: No data on PSP-related QoL or caregiver burden are available in France In addition, the factors determining these aspects of the disease are poorly understood. The motor handicap obviously reduces patients' QoL and increases the caregivers' burden. However the impact of the cognitive and behavioural disturbances and particularly the reduction of social interactions on the QoL of patients and caregiver burden have been less studied.

ELIGIBILITY:
Inclusion Criteria (patients)

Female or male, age ≥ 40 years at the time of onset of symptoms

* diagnosis of possible or probable PSP according to the criteria of Litvan (1996b)
* agreeing to participate in the study
* subject with no severe cognitive impairment (MMS> 20/30)
* subject who does not have psycho-behavioral comorbidity deemed to be severe enough to make his assessment impossible
* subject not presenting a measure of legal protection

Exclusion Criteria (patients)

* Age <40 years at the onset of symptoms
* Diagnosis other than PSP (including other Parkinsonian syndromes)
* Presence of another concomitant neurological disease
* subject with severe cognitive impairment (MMS≤20 / 30)
* subject presenting psycho-behavioral comorbidities considered sufficiently severe to make it impossible to evaluate
* subject under legal protection
* subject not affiliated to a social security scheme

Inclusion Criteria (caregivers)

* Female or male, age ≥ 18 years
* designated by the patient as the person closest to him / her
* agreeing to participate in the study
* subject affiliated to a social security scheme

Exclusion Criteria (caregivers)

* Age <18 years
* Not designated by the patient as the person closest to him / her
* Not agreeing to participate in the study
* subject not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PSP patients with their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
score of PSP-QoL questionnaire | 1 hour
  the score obtained by group will be compare
  Progressive Supranuclear Palsy (PSP) Quality of Life questionnaire by Schrag and collaborators in 2006.
  14 items, 5 degree from no problem, slight problem, moderate problem, marked problem to extreme problem (1 to 5 points) minimum score:14 maximum score : 70

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France